CLINICAL TRIAL: NCT04591522
Title: The Study of HIF-1α in Cirrhosis by Fecal Microbiota Transplantation
Brief Title: Fecal Microbiota Transplantation in Cirrhosis
Acronym: FMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yongping_Chen
Record Dates: First submitted 2020-08-25; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-08

CONDITIONS: Cirrhosis, Liver
Keywords: Cirrhosis；fecal Microbiota Transplantation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT group (Experimental): Patients were carried by fecal microbiota transplantation which described in detail that fecal bacteria are extracted from the faeces of healthy people and poured into the intestines of patients.
  Interventions: Other: Healthy fecal bacteria liquid
- control group (No Intervention)

INTERVENTIONS:
Other: Healthy fecal bacteria liquid — Fecal bacteria liquid were obtained from healthy people by a feces processor, and perfused into the patient's intestine.
  Arms: FMT group

SUMMARY:
Patients with cirrhosis were recruitted and divided into cintrol group and FMT group. Patients in FMT group were carried by fecal microbiota transplantation, and biochemical indexes, intestinal flora and intestinal HIF expression were observed before and after FMT respectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cirrhotic
* aged 18-80 years.
* must be able to cooperate with treatment

Exclusion Criteria:

* Patients with severe cardiac, pulmonary and renal dysfunction;
* Patients with severe hypertension and cerebrovascular accidents;
* Patients with liver cancer or active infection are in the active stage of hepatic encephalopathy or gastrointestinal bleeding;
* Prothrombin activity ≤40%, platelet count < 50*10^9/L;
* Patients with intellectual and language disorders and mental disorders;
* Probiotics with antibiotic and drug grade were used within 3 months prior to sampling;
* There are prehepatic or posthepatic portal hypertension reasons;
* Drug history: anticoagulant therapy, use of antiplatelet drugs, and current use of beta blockers, statins or interferon (IFN) treatment;
* Peptic colon examination contraindications, such as intestinal perforation, intestinal obstruction, etc.
* Other researchers believe that patients should not be included in the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
blood ammonia | Change from baseline blood ammonia at 12 months
  blood ammonia in umol/L
alanine aminotransferase | Change from baseline alanine aminotransferase at 12 months
  alanine aminotransferase in U/L
aspartate aminotransferase | Change from baseline aspartate aminotransferase at 12 months
  aspartate aminotransferase in U/L
gut microbiome | Change from baseline gut microbiome at 12 months
  16S RNA sequencing in gut microbiome
white blood cell | Change from baseline white blood cell at 12 months
  white blood cell in /L
hemoglobin | Change from baseline hemoglobin at 12 months
  hemoglobin in g/L
blood platelet | Change from baseline blood platelet at 12 months
  blood platelet in/L
albumin | Change from baseline albumin at 12 months
  albumin in g/L
blood glucose | Change from baseline blood glucose at 12 months
  blood glucose in mmol/L
Serum creatinine | Change from baseline serum creatinine at 12 months
  Serum creatinine in umol/L
direct bilirubin | Change from baseline direct bilirubin at 12 months
  direct bilirubin in umol/L
indirect bilirubin | Change from baseline indirect bilirubin at 12 months
  indirect bilirubin in umol/L
prothrombin time activity percentage | Change from baseline prothrombin time activity percentage at 12 months
  prothrombin time activity percentage in %
liver stiffness | Change from baseline liver stiffness at 12 months
  liver stiffness in Kpa

SECONDARY OUTCOMES:
Concentration of HIF-1α in intestine | Change from baseline HIF-1α expression in intestine at 12 months
  Concentration of HIF-1α expression in intestine by western blot

CONTACTS AND LOCATIONS:
Overall Officials: yongping Chen, Prof, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sung CM, Lin YF, Chen KF, Ke HM, Huang HY, Gong YN, Tsai WS, You JF, Lu MJ, Cheng HT, Lin CY, Kuo CJ, Tsai IJ, Hsieh SY. Predicting Clinical Outcomes of Cirrhosis Patients With Hepatic Encephalopathy From the Fecal Microbiome. Cell Mol Gastroenterol Hepatol. 2019;8(2):301-318.e2. doi: 10.1016/j.jcmgh.2019.04.008. Epub 2019 Apr 18. PMID 31004827